CLINICAL TRIAL: NCT05328934
Title: Toward Use of the Synergy-based SoftHand Pro for Activities of Daily Living by Persons With Transradial Limb Loss: A Multi-site Clinical Trial
Brief Title: SoftHand Comparison Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other); Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-005070
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Upper Extremity Injury; Upper Extremity Deformities, Congenital; Amputation, Traumatic; Amputation, Congenital
MeSH Terms: conditions — Arm Injuries; Upper Extremity Deformities, Congenital; Amputation, Traumatic; Amputation, Congenital

STUDY DESIGN:
Intervention Model Description: Crossover design with first intervention randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Initial Assignment: SoftHand Pro (Experimental): This arm of the crossover design will begin the trial using the SoftHand Pro.
  Interventions: Device: SoftHand Pro; Device: Ossur i-Limb
- Initial Assignment: Ossur i-Limb (Active Comparator): This arm of the crossover design will begin the trial using the i-Limb.
  Interventions: Device: SoftHand Pro; Device: Ossur i-Limb

INTERVENTIONS:
Device: SoftHand Pro — Performance assessments utilizing the SoftHand Pro over an 8-week period.
Device: Ossur i-Limb — Performance assessments utilizing the i-Limb over an 8-week period.

SUMMARY:
A trial to compare the performance of the SoftHand Pro (SHP) and Ossur i-Limb in people with transradial limb loss over an 8-week period.

DETAILED DESCRIPTION:
This study will measure improvements in outcomes obtained from laboratory testing of the SHP and i-Limb from baseline to after 8 weeks of daily use. A secondary analysis will incorporate the subjects' existing prosthetic hands. Finally, surveys and usage data collected through the SHP and i-Limb firmware during daily use will complement data the aforementioned outcomes to explore factors that may be related to differences in grasping and manipulation performance.

ELIGIBILITY:
Inclusion Criteria:

1. the individual can successfully use their prosthesis, list the components used and that their current prosthesis is fitting properly (by performing a tension analysis);
2. the individual had unilateral transradial limb loss more than 6 months before the clinical evaluation because, to use a myoelectric prosthesis, the residual limb volume needs to be stable;
3. the individual is a proficient owner of one or more common myoelectric prosthetic hands, such as the Sensor Hand Speed and Bebionic.

Exclusion Criteria:

1. individuals who have had transradial amputation for less than 6 months;
2. individuals who have been fit and trained to use a prosthesis but chose not to use one;
3. individuals who use the i-Limb Quantum myoelectric prosthesis;
4. symptomatic brachial plexopathy, cervical radiculopathy or polyneuropathy (observed);
5. orthopedic, joint degeneration (i.e., arthritis, self-reported) affecting the hand or cervical spine that severely limit upper limb function (observed);
6. visual problems that would interfere with the grasping;
7. co-existing central nervous system disease with symptoms that limit upper extremity function (e.g., multiple sclerosis, motor neuron disease, myasthenia gravis, Parkinson's disease, dystonia) revealed in medical history;
8. limited range of motion as assessed through range of motion testing;
9. inability to follow study instructions;
10. use of medications that might affect sensory and/or motor functions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Functional Ability [1] | 8 Weeks
  Change in upper extremity function, as measured by the Activities Measure for Upper Limb Amputees (AM-ULA). Participants complete 17 tasks, rated on task completion, speed of completion, movement quality, skillfulness of prosthesis use, and independence from the use of other assistive devices or adaptive environments with the prosthesis. The scale is 0 to 4, with a higher number representing higher performance in each category. Scores in each category are averaged for a Grade in each task. Grades for the 17 tasks are averaged and multiplied by 40 for a final score of 0 - 40, with a higher number representing higher overall function.

SECONDARY OUTCOMES:
Upper Extremity Functional Ability [2] | 8 Weeks
  Change in upper extremity function, as measured by the Action Research Arm Test (ARAT). Participants perform up to 19 tasks categorized by grasp, grip, pinch, and gross movement. The scale is 0 to 3, with a higher number representing higher performance in each category. Categories are scored separately.
Upper Extremity Manual Dexterity | 8 Weeks
  Change in upper extremity gross manual dexterity, as measured by the Box and Blocks test. Participants are tested in a timed transfer of blocks from one side of a box to another side over a low partition. A higher number of blocks successfully transferred during the timed episode represents a higher level of upper extremity manual dexterity.
Hand Motor Function | 8 Weeks
  Change in fine and gross motor hand function, as measured by the Jebsen-Taylor Hand Function Test. Participants are timed in seven activities of daily living closely involving use of the hand, with a lower number of seconds required to complete the task representing a higher level of motor hand function.
Occupational Performance | 8 Weeks
  Change in participants' perceived occupational performance, as measured by the Canadian Occupational Performance Measure (COPM). Participants choose up to 5 occupational performance problems; their perception of their own performance and their satisfaction with their performance regarding each problem is measured on a 1 to 10 scale, with higher scores representing higher performance and satisfaction. The difference in performance and satisfaction is calculated, and then the differences for all problems together are totaled and averaged, with the average divided by the number of problems establishing the final score for each performance and satisfaction. Higher averages represent better perceived performance and satisfaction.
Quality of Life | 8 Weeks
  Change in participants' perceived quality of life, as measured by the the World Health Organization Quality of Life Disabilities Module (WHOQOL-DIS). Participants answer qualitative questions regarding patient activities, independence, and overall quality of life on a 1 to 5 scale, with a higher number indicating a higher concurrence or frequency related to the item in question, and totaled for a score which categorizes patient quality of life.
Upper Extremity Function and Pain | 8 Weeks
  Change in participants' perceived levels of upper extremity physical function and symptoms, as measured by the Disabilities of the Arm, Shoulder, and Hand Score (QuickDASH). Participants rate their difficulty with examples of physical function and their severity of physical symptoms on a 1 to 5 scale, with higher values representing more severe difficulties and symptoms. The scores are combined in a calculation which results in an overall score, with higher scores representing more severe overall difficulties and symptoms.
Overall Functional Performance | 8 Weeks
  Change in participants' perceived functional performance, as measured by the Patient-Specific Functional Scale. Participants select 5 or more activities for which they perceive a problem, rating their own performance of that activity on a scale of 0 to 10, with higher values representing greater ability to perform the activity. The scores are totaled and divided by the number of tasks for an average score, with higher values representing better performance.
Prosthesis Overall Functional Utility | 8 Weeks
  Change in participants' perception of the utility of their currently-used prosthesis, as measured by the Orthotics Prosthetics Users Survey - Upper Extremity Functional Status (OPUS). Participants rate the prosthetic's ease of use for a variety of daily activities, 23 of which are scored, on a 0 to 4 scale, with higher values representing easier use. Scores are totaled and converted to a 0 to 92 scale, with higher overall scores representing better functional utility with the prosthesis.
Arm Pain | 8 Weeks
  Change in participants' levels of pain is measured for subjects who have pain due to brachial plexopathy or neuropathy. A visual analog pain scale (VAS) specific to the limb testing the experimental device will be administered prior to, and after, the clinical measures. The VAS scale is measured by the subject's own perspective by using a 0 to 10 scale, with zero indicating no pain and ten being intolerable pain. These baseline metrics will be compared with performance metrics obtained using the same tests delivered at the end of the daily-use period.

OTHER OUTCOMES:
Prosthesis User Preference | 8 Weeks
  Changes in participants' perception of the utility, functional performance, ergonomics, and ease of use of their currently-used prosthesis, as measured by a custom Active Use questionnaire. Participants rate the extent to which they agree to 12 to 14 statements (depending of which prosthesis) on a 1 to 10 scale, with higher ratings representing closer agreement. Individual statements are assessed separately (no overall score).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Santello, Ph.D., Principal Investigator — Arizona State University; Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No